CLINICAL TRIAL: NCT02410473
Title: Evaluation of Coagulation Testing in Patients Undergoing Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Juan Ibla, Cardiac Anesthesiologist, Boston Children's Hospital
Other Study IDs: P00016625
Record Dates: First submitted 2015-04-02; First posted 2015-04-07 (Estimated); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Congenital Heart Disease
Keywords: Congenital Heart Disease; Point-of-care coagulation monitoring
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Collect discarded blood from 4 routine blood samples. These will be obtained at 4 different time-points: 1. After induction of anesthesia and placement of arterial line, 2. After cardiopulmonary Bipass (CPB), 3 minutes after protamine administration, 3. At the end of the surgery, before transfer to CICU, 4. 24- 48 hrs post-surgery in the ICU.
  Collect two 5 mL of urine samples. One sample prior to CPB, as well as following CPB, from an routinely placed Foley catheter.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Discarded blood samples — Will utilize the discarded blood from routine clinical blood samples to evaluate the input of the newer technologies that helped for the diagnostic of coagulopathy.
Other: Discarded Urine Sample — Will utilized the discarded urine samples from the routinely placed Foley catheter to measure the indices of oxidative stress.

SUMMARY:
Neonates, children with single ventricle congenital heart disease, and those undergoing multiple complex cardiac surgeries are at high risk of increased perioperative blood loss, and blood product transfusions. In addition, some of these patients will present an increased risk of postoperative thromboembolic complications. For a long time, bleeding management has been based on the empiric administration of different blood products (e.g. platelet concentrates, cryoprecipitates, and/or activated factor VII), topical hemostatic agents, and surgical manipulation. Recently, the use of viscoelastic tests (e.g. thromboelastography (TEG) or thromboelastometry (ROTEM)) increased, and allowed a better assessment of perioperative coagulopathy, and a more 'rational' treatment of bleeding. While TEG and ROTEM record the viscoelastic properties of whole blood by measuring mechanical impedance and related changes during clot formation, T2MR, a miniaturized, magnetic resonance-based diagnostic platform, measures how water molecules react in the presence of magnetic fields to evaluate a broad range of hemostasis measurements. In this study, we will prospectively collect demographic data, surgical characteristics, the amount of perioperative bleeding and blood product transfusion, results of laboratory assays, and postoperative outcomes (30-day follow-up or until discharge), with the aim to assess our current practice, and develop an algorithm-based approach for the administration of targeted blood product and pro-coagulant therapies. Our goals are: the reduction of blood product utilization, the reduction of the incidence of massive bleeding and postoperative thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* Neonates and infant patients (0 -12 months of age) undergoing complex cardiac surgical procedures
* cardiac surgery patient > 12 months of age who has previously undergone 2 or more sternotomies

Exclusion Criteria:

* child in a moribund condition (American Society of Anesthesiology (ASA 5)
* children with a hematological and/or oncological disease
* Jehovah witnesses
* If the child is only undergoing a patent ductus arteriosus (PDA) ligation or other procedures not considered at risk for thrombosis and/or bleeding or they do not provide consent for enrollment (e.g. Ventricular Septal Defect repair)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Neonates and infants undergoing cardiac surgery with cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate newer technologies for coagulation diagnostics with the aim to standardize bleeding management in high risk cardiac patients | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Juan Ibla, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Brummel-Ziedins K, Undas A, Orfeo T, Gissel M, Butenas S, Zmudka K, Mann KG. Thrombin generation in acute coronary syndrome and stable coronary artery disease: dependence on plasma factor composition. J Thromb Haemost. 2008 Jan;6(1):104-10. doi: 10.1111/j.1538-7836.2007.02799.x. Epub 2007 Oct 15. PMID 17944993
- [Background] Eisses MJ, Chandler WL. Cardiopulmonary bypass parameters and hemostatic response to cardiopulmonary bypass in infants versus children. J Cardiothorac Vasc Anesth. 2008 Feb;22(1):53-9. doi: 10.1053/j.jvca.2007.06.006. Epub 2007 Aug 22. PMID 18249331
- [Background] Emani S, Zurakowski D, Baird CW, Pigula FA, Trenor C 3rd, Emani SM. Hypercoagulability markers predict thrombosis in single ventricle neonates undergoing cardiac surgery. Ann Thorac Surg. 2013 Aug;96(2):651-6. doi: 10.1016/j.athoracsur.2013.04.061. Epub 2013 Jun 26. PMID 23809731
- [Background] Fries D, Innerhofer P, Streif W, Schobersberger W, Margreiter J, Antretter H, Hormann C. Coagulation monitoring and management of anticoagulation during cardiac assist device support. Ann Thorac Surg. 2003 Nov;76(5):1593-7. doi: 10.1016/s0003-4975(03)01034-8. PMID 14602292
- [Background] Koestenberger M, Cvirn G, Nagel B, Rosenkranz A, Leschnik B, Gamillscheg A, Beitzke A, Muntean W. Thrombin generation determined by calibrated automated thrombography (CAT) in pediatric patients with congenital heart disease. Thromb Res. 2008;122(1):13-9. doi: 10.1016/j.thromres.2007.08.016. Epub 2007 Oct 3. PMID 17915295
- [Background] Livingston ER, Fisher CA, Bibidakis EJ, Pathak AS, Todd BA, Furukawa S, McClurken JB, Addonizio VP, Jeevanandam V. Increased activation of the coagulation and fibrinolytic systems leads to hemorrhagic complications during left ventricular assist implantation. Circulation. 1996 Nov 1;94(9 Suppl):II227-34. PMID 8901751
- [Background] Nankervis CA, Preston TJ, Dysart KC, Wilkinson WD, Chicoine LG, Welty SE, Nelin LD. Assessing heparin dosing in neonates on venoarterial extracorporeal membrane oxygenation. ASAIO J. 2007 Jan-Feb;53(1):111-4. doi: 10.1097/01.mat.0000247777.65764.b3. PMID 17237658
- [Background] Tappenden KA, Gallimore MJ, Evans G, Mackie IJ, Jones DW. Thrombin generation: a comparison of assays using platelet-poor and -rich plasma and whole blood samples from healthy controls and patients with a history of venous thromboembolism. Br J Haematol. 2007 Oct;139(1):106-12. doi: 10.1111/j.1365-2141.2007.06732.x. PMID 17854314
- [Background] Vittinghoff E, McCulloch CE. Relaxing the rule of ten events per variable in logistic and Cox regression. Am J Epidemiol. 2007 Mar 15;165(6):710-8. doi: 10.1093/aje/kwk052. Epub 2006 Dec 20. PMID 17182981